CLINICAL TRIAL: NCT01805700
Title: Effects of Acute Intake of Caffeine Enhanced Energy Drinks on Blood Glucose, Some Physiological Parameters and Cognitive Performance in Patients With Type 1 Diabetes
Brief Title: Effects of Acute Intake of Caffeinated Beverages in Type 1 Diabetes
Acronym: REDBULL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: B091217
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1; diabetes; caffeine-enhanced energy drink; cardiac output; glucose; cognitive performance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regular caffeine enhanced energy drink (Experimental): Regular caffeine enhanced energy drink (containing 240mg caffeine & 84g glucose) e.g. regular red bull cans (x3)
  Interventions: Other: Caffeine enhanced energy drink
- Diet Caffeine enhanced energy drink (Experimental): Diet Caffeine enhanced energy drink ( containing 240mg of caffeine alone) e.g. Red Bull light)
  Interventions: Other: Caffeine enhanced energy drink
- Glucose drink (Active Comparator): Glucose drink (containing 84g glucose alone)
  Interventions: Other: Glucose drink

INTERVENTIONS:
Other: Caffeine enhanced energy drink — Comparison of different energy drinks
  Other Names: Red Bull
  Arms: Diet Caffeine enhanced energy drink; Regular caffeine enhanced energy drink
Other: Glucose drink — Glucose drink (containing 84mg glucose alone)
  Arms: Glucose drink

SUMMARY:
The aim of this pilot study is to determine the impact of caffeine-enhanced energy drinks on blood glucose excursion on heart rate, blood pressure, cardiac output and cognitive performance in patients with type 1 diabetes.

Knowledge acquired may inform a wider study of the impact of these drinks.

This is a randomised, cross over blinded study in which all participants will participate in the 3 arms of the study.

The study will consist of 3 phases, each lasting 3 days. A different study drink will be administered during each phase. There will be an initial screening visit and a pre- study visit before each study phase. Each participant will make 10 visits to the research centre.

There will be a week wash out period between each study phase. Prior to each study phase, there will be a 3 day caffeine and alcohol abstinence run-in period.

Study drinks will be matched for taste and volume (as far as possible) and will be administered by the use of opaque cups, lids and straws to enable double-blind randomisation for both researcher and participants. Administration of the study drink to participants will be based on Latin squares to provide a balanced treatment order.

During the 3 days study period; participants will be required to abstain from all other caffeine containing beverages or confectioneries.

The secondary aim is to determine if tolerance to cardiovascular effects of caffeine-enhanced energy drinks is developed following acute short term ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥18 years
* Confirmed diagnosis of Type 1 diabetes of more than one year duration
* Participants who use multiple daily injections of basal and meal-time analogue insulin.
* Ability to perform daily finger stick measurements of blood glucose levels
* Adequate contraceptive control
* Provision of informed consent

Exclusion Criteria:

* Hypoglycaemia unawareness
* Coronary heart disease
* Cardiac arrhythmia
* Structural heart lesions,
* Autonomic neuropathy
* Psychiatry illness,
* Epilepsy
* Migraine
* Caffeine intolerance
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose level in all patients as a measure of tolerability | Day 1, Day 2 and Day 3

SECONDARY OUTCOMES:
The effects on certain mood states, e.g. energetic arousal, tense arousal and hedonic tone following the consumption of caffeinated energy drinks in comparison with caffeine free glucose in patients with type 1 diabetes | Day 1, day 2 and day 3
Changes in reaction time and digit symbol substitution test score | Day 1, day 2 and day 3
Changes in heart rate, systolic and diastolic blood pressure in all patients. | Day 1, day 2 and day 3

CONTACTS AND LOCATIONS:
Overall Officials: Tolulope Olateju, MRCP, Principal Investigator — The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Locations (1):
- The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, Dorset, United Kingdom